CLINICAL TRIAL: NCT07020585
Title: 2024 National Survey of Early Care and Education (NSECE) Longitudinal Follow-ups
Status: Active, not recruiting | Type: Observational
Sponsor: National Opinion Research Center (Other)
Collaborators: Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rupa Datta, Distinguished Senior Fellow, National Opinion Research Center
Other Study IDs: HHSP233201500048I-FU
Record Dates: First submitted 2025-05-29; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Children Under 13
Keywords: Early care and education; Center-based providers; Home-based providers; Caregivers; Child care; Workforce; ECE

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Households: Interviews conducted with households (1) with incomes under 300% of the federal poverty (FPL) and with at least one resident child under the age of 13 years and/or (2) who had used paid care by an individual in the spring of 2024. Households will be drawn from the 2024 NSECE.
- Workforce (Classroom Staff): Interviews conducted with individuals who were employed in 2024 in center-based ECE programs working directly with children in classrooms serving children age 5 years and under, not yet in kindergarten. Participants will be drawn from the 2024 NSECE.

SUMMARY:
The National Survey of Early Care and Education (NSECE) captures families' needs, preferences, and choices of non-parental care for children under age 13 and providers' child care and early education offerings. Since the NSECE was conducted in 2019, the landscape of ECE has changed dramatically. Funding for early childhood programming has grown as policymakers recognize the important role access to ECE plays for families as a work support for parents and an investment in children's future educational and economic opportunities. At the same time, beginning in 2020, the nation experienced the COVID-19 pandemic, leading to significant shifts in the U.S. economy. These circumstances likely altered parents' use of ECE and the labor market and economic forces in which ECE providers operate. The 2024 NSECE builds on findings from the 2012 and 2019 NSECE to allow for comparisons of supply and demand of child care and early education over the 12 years that span data collection.

The 2024 NSECE Follow-up studies build on findings from the 2024 NSECE to allow for more in-depth information on how families search for and select care for their children, as well as an understanding of workforce career trajectories. The 2024 NSECE Follow-up studies aim to inform future policy discussions about child care and early education at the local, state, and national levels by providing data to:

* Build on the data collected in 2024 to collect additional and more in-depth data.
* Capture how low-income households learn about and make use of financial assistance in seeking and selecting ECE, with additional focus on paid individual care arrangements.
* Document patterns of retention and attrition among individuals in the center based ECE workforce.

DETAILED DESCRIPTION:
To expand on the 2024 NSECE data regarding the use of ECE, the NSECE Follow-up is conducting two nationally representative surveys. These surveys target (1) households and (2) center-based provider workforce to gather more detailed information.

The Household Survey is being conducted with households participating in the 2024 NSECE and either a. reporting a paid individual ECE arrangement in the 2024 NSECE, and/or b. having at least one resident child under age 13 and who reported incomes under the 300% Federal poverty level in the 2024 NSECE. These two populations are not mutually exclusive. Eligible respondents are identified by the information collected on 2024 NSECE. This survey documents the ECE search and selection experiences of households with low incomes. Key questionnaire topics include details on households' awareness of and experience with publicly-funded ECE programs, how households selected ECE arrangements for fall 2024, who provided paid individual care to the households' children in early 2024, whether households sought financial assistance for ECE, and the current status of individual care arrangements used in spring 2024.

These data will help to answer such research questions as (1) Which arrangements from winter/spring 2024 are still in effect in fall 2024? (2) What ECE programs are families aware of in their local area, and how much do they know about program rules and the family's own eligibility? (3) What factors contribute to how a family undertakes search and selection for their children? (4) Which desired characteristics of providers are most challenging for parents to satisfy in their search activities? (5) What steps did families take to find affordable care? The Workforce (Classroom Staff) Survey sample is comprised of individuals who participated in the 2024 NSECE Workforce Survey (i.e., served as center-based classroom-assigned instructional staff in 2024). This survey documents the career trajectory of ECE classroom staff, identifying individuals who still work at the same center, individuals who moved to a different center but still work in ECE, individuals who do not currently work in ECE, and individuals who do not currently work.

The questionnaire identifies patterns of retention and attrition among individuals in the center based ECE workforce. Key questionnaire topics include identifying job transitions, their current role for the individuals who are in the working force, career trajectories, and more information about their current job.

The data will answer such questions as (1) What are the characteristics and experiences of educators who leave an ECE classroom role? (2) What reasons do workers report for leaving their classroom roles? What center, classroom, or worker characteristics are associated with workers leaving classroom roles? (3) What motivates educators to stay in their current centers and in ECE? (4) What community, center, professional or personal characteristics are related to advancement or improvements in compensation over that period? (5) Which educators have looked for other employment recently? (6) What do educators report about their job satisfaction?

ELIGIBILITY:
Inclusion Criteria:

* Households which participated in 2024 NSECE (1) with incomes under 300% of the federal poverty (FPL) and with at least one resident child under the age of 13-years and/or (2) who had used paid care by an individual in the spring of 2024
* Respondents for the workforce (classroom staff) survey are selected from the 2024 NSECE respondents and were employed in early 2024 in center-based ECE programs working directly with children in classrooms serving children age 5 years and under, not yet in kindergarten.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Households that participated in 2024 NSECE Household Survey. Households with children under 13 years.
  Individuals who participated in the 2024 NSECE Workforce (Classroom Staff) Survey working in center-based classrooms.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Search and Selection of ECE | January 2025 to May 2025
  The household questionnaire collects information on how each household seek and choose ECE, including information about the status of ECE arrangements from the main interview, if and how households seek financial assistance for ECE, and the origin and current status of individual care arrangements used in 2024.
Career Trajectories of ECE Workforce | September 2025 to December 2025
  The workforce classroom staff questionnaire collects information about job transition (current employment status, current role, including occupation, work schedule, recent job search), career trajectories (career experiences in different ECE settings, wage and role progression, non-ECE career experience), current employment characteristics (compensation, current work location, work environment, job satisfaction), and current work in ECE (current title, characteristics of current position, program characteristics, wellness support, experiences of program turnover, and promotions).

CONTACTS AND LOCATIONS:
Overall Officials: Rupa Datta, PhD, Principal Investigator — NORC at the University of Chicago
Locations (1):
- NORC at the University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No